CLINICAL TRIAL: NCT06457841
Title: Black Adult Resilience Study
Brief Title: Stress and Resilience
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Priscilla Lui, Associate Professor, Department of Psychology, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: STUDY00018058; R01DA058626 (NIH)
Record Dates: First submitted 2024-05-28; First posted 2024-06-13 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Alcohol Use; Cannabis Use
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Direct Interpersonal Exchange (Experimental): Simulated a negative personally relevant interpersonal experience that is received directly from a perpetrator, commonly experienced in everyday lives
  Interventions: Behavioral: Direct Interpersonal Exchange
- Vicarious Interpersonal Exchange (Experimental): Hearing or observing a negative personally relevant interpersonal experience that is reported by another person of the same background
  Interventions: Behavioral: Vicarious Interpersonal Exchange
- Daily Hassles (Placebo Comparator): Day-to-day stressors associated with school, work, finances
  Interventions: Behavioral: Daily Hassles

INTERVENTIONS:
Behavioral: Direct Interpersonal Exchange — Simulated a negative personally relevant interpersonal experience that is received directly from a perpetrator, commonly experienced in everyday lives
  Arms: Direct Interpersonal Exchange
Behavioral: Vicarious Interpersonal Exchange — Hearing or observing a negative personally relevant interpersonal experience that is reported by another person of the same background
  Arms: Vicarious Interpersonal Exchange
Behavioral: Daily Hassles — Day-to-day stressors associated with school, work, finances
  Arms: Daily Hassles

SUMMARY:
Alcohol and cannabis are the most misused psychoactive substances in the United States. The proposed research examines how personally relevant stressful experiences may lead to alcohol and cannabis use. The proposed research is also designed to identify possible targets for prevention and treatment efforts to help reduce drug use.

ELIGIBILITY:
Inclusion Criteria:

* Of Afro-descent
* Proficient in English
* Alcohol and/or cannabis use at least 2-3 times in the past month
* Endorse having used alcohol and/or cannabis to cope

Exclusion Criteria:

* Having participated in similar studies by the research team
* Obtain cut-off scores on scale items indicating possible loss of control and needing to cut down or quit alcohol and/or cannabis use
* In or seeking treatment for alcohol and/or cannabis use disorder

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 456 (Estimated)
Dates: Start 2024-05-09 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Momentary Alcohol and/or Cannabis Craving | Immediately after the intervention (i.e., within 1 minute)
  Momentary Alcohol and Cannabis Craving Scale will be administered (adapted from the Momentary Cannabis Craving Scale; Davis et al., 2024) immediately after the intervention. Mean scores will range from 1 to 7, with higher scores indicating greater momentary craving.
Duration of Alcohol and Cannabis Intoxication | 48 Hours Post-Intervention
  Self-reported number of hours of intoxication within 48 hours after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: P. Priscilla Lui, Ph.D., Principal Investigator — University of Washington
Locations (2):
- United States (2):
  - Southern Methodist University, Dallas, Texas
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No